CLINICAL TRIAL: NCT05794945
Title: OPTIMISTOptimizing Mastitis Identification and Treatment
Brief Title: Optimizing Mastitis Identification and Treatment
Acronym: OPTIMIST
Status: Recruiting | Type: Observational
Sponsor: University of Tromso (Other)
Collaborators: Norwegian Institute of Public Health (Other Government); The University of Western Australia (Other); Helse Nord (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023/578416 (REK)
Record Dates: First submitted 2023-02-24; First posted 2023-04-03 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Mastitis Postpartum
Keywords: Breast inflammation; Clinical mastitis; Sub-clinical mastitis
MeSH Terms: conditions — Mastitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Researchers will collect human milk samples and skin swabs. Samples will be used for culture dependent assessment of the microbiological composition in milk and on breast skin and breast nipple.
  Researchers will isolate microbial DNA in order to perform whole genome sequencing and amplicon sequencing to map the microbial community in breastmilk.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breastfeeding mothers: In this study breastfeeding mothers will be included. Samples will be collected from breast-feeding mothers experiencing mastitis Samples will be collected from breast-feeding mothers after the mastitis episode is resolved Breastfeeding mothers will be sampled at each mastitis episode, and with the final sample collected after a maximum of 12 months

SUMMARY:
The goal of this observational study is to gain more information about the aetiology and progression of mastitis and breast inflammation, in order to develop evidence-based clinical guidelines and treatment plans, especially concerning judicious use of antibiotics.

The main questions it aims to answer are:

* Do clinical symptoms differ between inflammatory and infectious mastitis?
* What is the microbial composition in human milk, and does it change before, during, and after episodes of mastitis?
* Does the bacterial composition change due to antibiotic treatment?
* Are all mastitis episodes treated with antibiotics bacterial mastitis?
* Do mothers with recurrent mastitis have a distinct microbial composition?
* Are there immunological markers that can differentiate between bacterial and inflammatory mastitis?

Researchers will compare breastfeeding women with and without mastitis to see if the microbiological composition in milk and on the skin of the breast and breast nipple differs.

DETAILED DESCRIPTION:
Mastitis (breast inflammation) is experienced by up to one-fifth of all breastfeeding mothers. Mastitis is a painful condition and a leading cause of early weaning, an undesired outcome with potentially negative implications for both mother and baby. Empirical evidence explaining the aetiology of mastitis is lacking; thus the definitions and treatment of mastitis is conflicting. The recent mechanobiological model proposes that the mechanical forces of lactation, especially at the onset of milk production, can cause damage to the mammary tissue, which induces an inflammatory response. Concurrently a growing amount of evidence shows that bacteria previously written off as contaminants have a role in mastitis which has been overlooked. The dynamics between the mechanobiological model and bacterial colonization have not yet been investigated. To fill this knowledge gap, researchers will conduct a longitudinal study collecting milk samples and questionnaires during the breastfeeding period with a particular emphasis on mastitis. Milk and skin swab samples will be used for culture dependent and culture independent assessment of the microbial composition in mastitis, and will be compared to the composition found in mothers without mastitis.

The main objective of this clinical study is to gather empirical data to provide an evidence-based update to the clinical guidelines for mastitis diagnosis and care. This will provide a foundation for improving the treatment and prevention of mastitis, with better outcomes for mothers and newborns.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant mothers aged > 18
* mothers must understand information given in Norwegian or English
* participants must be willing to complete study questionnaires
* participants must be willing to and provide biological samples

Exclusion Criteria:

* No exclusion criteria

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — This study will include breastfeeding mothers
Study Population: Pregnant mothers aged > 18 years planning to give birth at University Hospital Noth Norway (UNN), with the intention to breastfeed and with an address in Tromsø municipality.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Determination of the microbial composition in human milk from mothers without mastitis by MALDTI-TOF and Illumina sequencing | 18 months
  In order to investigate if there is a particular microbial composition of the human milk that leads to mastitis, the microbial composition in human milk from mothers without mastitis will be assessed. The investigators will collect milk samples from all enrolled mothers at day 6-7 after birth. Milk samples will be stored at -20 until further processing.
  Mothers who develop mastitis will be further sampled as described in outcome 2. Samples will be analyzed using culture dependent and culture independent methods. Following culturing of the milk samples, colonies will be analysed by Matrix-assisted laser desorption/ionization-time of flight (MALDI-TOF) to identify bacterial species. DNA will be isolated from the same milk sample.16S rRNA amplicon sequencing of DNA from milk samples will be performed using the Illumina technology, in order to get an overview of the total bacterial composition.
Determination of the microbial composition in human milk from mothers at onset of mastitis by MALDTI-TOF and Illumina sequencing | 18 months
  The investigators will investigate if the microbial composition in human milk changes at onset of mastitis. By analysing possible changes in microbial composition the investigators will assess if the mastitis symptoms are caused by microorganisms, or if the symptoms of mastitis are inflammatory. Milk samples will be collected by the mother at onset of mastitis, 24 hours after onset of symptoms and after resolution of symptoms. If the mastitis episode is treated with antibiotics, a new sample will be taken 24 hours after cessation of antibiotic treatment. Milk samples will be stored at -20 until further processing. Samples will be analyzed using culture dependent, and culture independent methods. Following culturing of the samples, colonies will be analysed by MALDI-TOF to identify bacterial species. 16S rRNA amplicon sequencing of DNA from milk samples will be performed using the Illumina technology, in order to get an overview of the total bacterial composition.
Assessment of the microbial composition on nipples of mothers without mastitis | 18 months
  It is no agreement on if mastitis causing bacteria originate from the breast nipple, or if they are part of the milk microbiome. We will sample the breast nipples in order to investigate if microorganisms colonizing the breast skin enter the mammary glands, and potentially cause mastitis. A skin swab of the nipple (both breasts) will be taken at day 6-7 after birth. Following culturing of the swab, bacterial colonies will be analysed by MALDI-TOF to identify bacterial species. The skin swabs will be collected at the same timepoints as collection of milk samples.
Assessment of the microbial composition on nipples of mothers with mastitis | 18 months
  It is no agreement on if mastitis causing bacteria originate from breast nipple, or if they are part of the milk microbiome. We will sample the breast nipples in order to investigate if microorganisms colonizing the breast skin enter the mammary glands, and potentially cause mastitis.
  When the mother experiences symptoms of mastitis the mother will collect a skin swab sample. Following culturing of the swab, bacterial colonies will be analysed by MALDI-TOF to identify bacterial species. The skin swabs will be collected at the same timepoints as collection of milk samples.The microbial composition on nipples of mothers with mastitis will also be compared to the nipple microflora of mothers without mastitis in order to see if there is a correlation between particular skin colonizing bacteria that cause mastitis.
The concentration of immunological markers in milk from mothers without mastitis | 18 months
  A milk sample will be collected at day 6-7 after birth, and the concentration of immunological markers will be assessed in the milk of mothers without mastitis. The concentration (pg/ml) of 8 immune factors, including innate immune factors (IL6, IFNγ, TNFα), acquired immune factors (IL2, IL4, IL10), chemokines (IL8), and growth factor (GMCSF), will be determined by magnetic bead-based multi- plex immunoassays, using a Bioplex 200 instrument (Bio-Rad, Hercules, CA, USA).
The concentration of immunological markers in milk from mothers with mastitis | 18 months
  In order to determine if there is an increase in the immunological markers present in milk from mothers with mastitis, milk samples will be collected at onset of mastitis symptoms and 24 hours after cessation of symptoms. If the mother requires antibiotic treatment , samples will be collected at onset of treatment and 24 hours after cessation of antibiotic treatment. The concentration (pg/ml) of 8 immune factors, including innate immune factors (IL6, IFNγ, TNFα), acquired immune factors (IL2, IL4, IL10), chemokines (IL8), and growth factor (GMCSF), will be determined by magnetic bead-based multi- plex immunoassays, using a Bioplex 200 instrument (Bio-Rad, Hercules, CA, USA).The investigators will assess if the concentration of immunological markers differs in bacterial mastitis and inflammatory mastitis.
Mapping of mastitis symptoms by detailed Questionnaires | 18 months
  The mothers will be asked to fill in a detailed questionnaire regarding breastfeeding practice and symptoms of mastitis.
  The questionnaire will accompany the collection of milk samples as described in outcome 1and 2.

CONTACTS AND LOCATIONS:
Overall Officials: Jorunn Pauline Cavanagh, PhD, Principal Investigator — The Arctic university of Norway-UiT
Locations (2):
- Norway (2):
  - Tromsø municipality, health centre, Tromsø, Troms
  - UiT-The Arctic University of Norway, Tromsø

IPD SHARING:
Plan to Share IPD: Yes
Researchers will share questionnaires, Informed consent forms and protocol, after data is published.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available after publication
Access Criteria: Access upon request

REFERENCES:
- [Result] Wilson E, Woodd SL, Benova L. Incidence of and Risk Factors for Lactational Mastitis: A Systematic Review. J Hum Lact. 2020 Nov;36(4):673-686. doi: 10.1177/0890334420907898. Epub 2020 Apr 14. PMID 32286139
- [Result] Mitchell KB, Johnson HM, Rodriguez JM, Eglash A, Scherzinger C, Zakarija-Grkovic I, Cash KW, Berens P, Miller B; Academy of Breastfeeding Medicine. Academy of Breastfeeding Medicine Clinical Protocol #36: The Mastitis Spectrum, Revised 2022. Breastfeed Med. 2022 May;17(5):360-376. doi: 10.1089/bfm.2022.29207.kbm. PMID 35576513
- [Result] Grzeskowiak LE, Saha MR, Ingman WV, Nordeng H, Ystrom E, Amir LH. Incidence, antibiotic treatment and outcomes of lactational mastitis: Findings from The Norwegian Mother, Father and Child Cohort Study (MoBa). Paediatr Perinat Epidemiol. 2022 Mar;36(2):254-263. doi: 10.1111/ppe.12824. Epub 2021 Nov 28. PMID 34841537
- [Result] Castro I, Garcia-Carral C, Furst A, Khwajazada S, Garcia J, Arroyo R, Ruiz L, Rodriguez JM, Bode L, Fernandez L. Interactions between human milk oligosaccharides, microbiota and immune factors in milk of women with and without mastitis. Sci Rep. 2022 Jan 25;12(1):1367. doi: 10.1038/s41598-022-05250-7. PMID 35079053